CLINICAL TRIAL: NCT06130358
Title: HeART-BRAIN : Investigating the Effects of a Museum Intervention on the Psychological and Cardiac Health of Older Adults With and Without Atrial Fibrillation
Brief Title: Investigating the Effects of a Museum Intervention on the Psychological and Cardiac Health of Older Adults
Acronym: HeART-BRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Louis Bherer (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Université de Montréal (Other); Mitacs (Industry)
Responsible Party: Sponsor-Investigator, Louis Bherer, Direction of EPIC Center, Montreal heart Institute, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ICM 2024-3325
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation Recurrent; Aging
Keywords: Museum visits; Neurocognition; Stress; Cardiovascular functioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Well-Being Museum intervention (Experimental): The well-being intervention comprises six weeks of weekly museum visits, performed in groups of 10 participants. The well-being approach is based on the support of a museum mediator. His role is to help visitors to develop a more personal and sensitive understanding of artworks. To do this, he encourages the expression of feelings, impressions, and interpretations of the artwork, and supports exchanges within the group of visitors. With the mediator's support, the participants should be able to adopt a more subjective approach to the artwork, favoring their engagement when contemplating it.
  Interventions: Other: Experimental: Well-being intervention followed by classic intervention; Other: Experimental: Classic intervention followed by well-being intervention
- Classic Museum intervention (Active Comparator): The classic intervention comprises six weeks of weekly museum visits, performed in groups of 10 participants. The classic museum session will be performed according to what is typically provided to visitors as part of a guided visit to the museum. Each visit will be accompanied by a volunteer guide trained in art history. He will guide participants across artworks and provide information about art pieces, the artist, and the historical context. The volunteer guide will provide context and informative content about the artwork without intending to influence the discussions and the visitor's apprehension of the artwork.
  Interventions: Other: Experimental: Well-being intervention followed by classic intervention; Other: Experimental: Classic intervention followed by well-being intervention

INTERVENTIONS:
Other: Experimental: Well-being intervention followed by classic intervention — 2 x 6 weeks of weekly museum visits
Other: Experimental: Classic intervention followed by well-being intervention — 2 x 6 weeks of weekly museum visits

SUMMARY:
In a recent report, the World Organization for Health provided some evidence that artistic and cultural activities can support the health and well-being of the population. Our previous research suggests that the effect of museum visits on well-being and stress might be tied to relaxing proprieties of contact with art objects, especially when the artwork is viewed with an introspective and self-reflexive approach. This study addresses the effect of a well-being museum intervention of six weeks on cerebral activity associated with artwork contemplation during a museum visit and assesses how it affects the psychological and cardiovascular health of older adults with and without atrial fibrillation. The well-being intervention will engage the participant in a series of 6 visits, in groups of 10, oriented on his feelings, impressions, and interpretations of artworks. This well-being museum intervention will be compared to visits typically provided in the museum, in a cross-over single-blinded design.

ELIGIBILITY:
Inclusion Criteria:

* Men/women aged 50 and over,
* Presenting normal or corrected vision and hearing,
* With or without controlled Atrial fibrillation,
* No specific expertise in visual arts (official degree or training relating to the visual arts),
* Occasionally attended museums and exhibitions (≤ 6 times per year).

Exclusion Criteria:

* Score > 5/15 on the geriatric depression scale,
* Score on the telephone version of the MMSE < 19,
* Psychiatric or neurological diagnosis,
* Presence of major functional limitations likely to affect the individual's ability to stand and walk independently.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in the activity evoked within the ventrolateral prefrontal cortex during the contemplation of artwork | Before and after the 6 weeks of interventions
  Hemodynamic variations in the region of interest (concentration of oxygenated hemoglobin [HbO2], no units).

SECONDARY OUTCOMES:
Change in the activity evoked within the medial prefrontal cortex during the contemplation of artwork | Before and after the 6 weeks of interventions
  Hemodynamic variations in the region of interest (concentration of oxygenated hemoglobin [HbO2], no units).

OTHER OUTCOMES:
Change in Heart rate | Before and after the 6 weeks of interventions
  bpm
Change in arterial pressure | Before and after the 6 weeks of interventions
  mmHg
Change in salivary cortisol concentration | Before and after the 6 weeks of interventions
  microg/l
Change in emotionnal regulation | Before and after the 6 weeks of interventions
  Difficulties in Emotion Regulation Scale DERS-F scale (Score ranges from 36-180, with a higher score indicating more emotion regulation problems)
Change in perceived stress | Before and after the 6 weeks of interventions
  Perceived Stress Scale questionnaire (Score ranges from 0-4, with 0 no stress,1 mild stress, 3 moderate stress and 4 severe).
Change in Depressive symptomatology | Before and after the 6 weeks of interventions
  Geriatric Depression Scale questionnaire (Score ranges from 0-30, with a higher score indicating larger depressive symptomatology).
Change in Quality-of-life | Before and after the 6 weeks of interventions
  36-Item Short Form Health Survey (Scale ranges from 0-100, with a higher score indicating a better health status).
Change in Perceived social support | Before and after the 6 weeks of interventions
  Lubben Social Network Scale questionnaire (Score ranges from 0-30, with a higher score indicating more social engagement).
Change in Repetitive negative thinking | Before and after the 6 weeks of interventions
  Perseverative thinking questionnaire (Score ranges from 0-60, with a higher score indicating more repetitive negative thinking).
Change in perceived fatigue | Before and after the 6 weeks of interventions
  Fatigue Severity Scale (Score ranges from 9-63, with a higher score more fatigue)
Change in global cognition | Before and after the 6 weeks of interventions
  MoCA total score (Score ranges from 0-30, with a higher score indicating better performance)
Change in executive functioning | Before and after the 6 weeks of interventions
  Computerized Stroop task, Reaction time (ms)
Self-reported masculinity and femininity trait | Baseline
  Short Form Bem Sex-Role Inventory questionnaire (30 items questionnaire with 10 items assessing the femininity traits, 10 items assessing the masculinity traits, and 10 items neutral, not scored. Two scores are calculated for femininity and masculinity, respectively, and range from 10-70, whit a higher score indicating a higher femininity or masculinity trait).
Cognitive Reserve | Baseline
  Rami and colleagues' cognitive reserve questionnaire (Scale ranges from 0-26, with a higher score indicating a greater cognitive reserve).

CONTACTS AND LOCATIONS:
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No